CLINICAL TRIAL: NCT02418416
Title: Calcium Ionophore Together With Strontium Chloride Would Likely Have a Positive But Non-traumatic Impact on Human Embryo Development
Brief Title: Novel Approach With Double Agent Artificial Oocyte Activation for Repeated Fertilization Failure Due to Combined Sperm and Oocyte Factor
Acronym: CISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Al Baraka Fertility Hospital (Other); Banon IVF Center Assiut, Egypt (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Laboratory Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IbnSina Hospital IVF
Record Dates: First submitted 2015-04-06; First posted 2015-04-16 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double activation (Experimental): The Oocytes in this arm will undergo double activation with Ca ionophore 5 micro mol for 20 min them Strontium chloride 10 micro mol for 60 min.
  Interventions: Other: Oocyte double chemical activation
- Control arm (No Intervention): The Oocytes will undergo Intracytoplasmic sperm injection only

INTERVENTIONS:
Other: Oocyte double chemical activation — Oocyte double chemical activation
  Arms: Double activation

SUMMARY:
Novel approach for Oocyte fertilization failure for difficult cases not respond to traditional methods of assisted reproduction as intracytoplasmic sperm injection.

DETAILED DESCRIPTION:
In some cases undergoes assisted reproduction technique specially Intracytoplasmic sperm injection, in subgroup of patient they fail to fertilize or poorly fertilized, some authors recommend chemical activation for those group of patient with Ca ionophore but still with Ca ionophore there are some cases with total fertilization failure or low fertilization specially in those patient with 2 separate factors like teratozoospermia with poor quality Oocytes so the investigators decided to test the effect of double activation methods by using tow agents proven with life birth rate Ca ionophore and strontium chloride.

We Do intracytoplasmic sperm injection and immediately activate oocyte with Ca Ionophore followed by strontium chloride activation and monitoring the embryogenesis until the blastocyst formation and pregnancy outcome in multicenter assessment.

ELIGIBILITY:
Inclusion Criteria:

* poor sperm
* poor quality Oocytes
* previous failed fertilization
* previous poor embryogenesis

Exclusion Criteria:

* normal patient
* previous successful outcome

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy rate ( % ) | 3 months
  To predict percentage of pregnant women from those will undergo Embryo transfer

SECONDARY OUTCOMES:
Blastocyst rate ( % ) | 3 months
  Number of embryos will reach blastocyst stage at day 5 post Intracytoplasmic sperm injection

CONTACTS AND LOCATIONS:
Locations (3):
- Al Barka fertility center, Bahrain, Bahrain
- Egypt (2):
  - Banon fertility center, Asyut
  - IbnSina IVF unit, IbnSina Hospital, El Areef Square, Sohag